CLINICAL TRIAL: NCT02253329
Title: The Effect of Neuromuscular Electrical Stimulation on Post-prandial Protein Accretion During the Day and Prior to Sleep
Brief Title: NMES During the Day and Prior to Sleep
Acronym: ESPRO2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MEC 14-3-042
Record Dates: First submitted 2014-09-29; First posted 2014-10-01 (Estimated); Last update posted 2015-05-21 (Estimated); Status verified 2015-05

CONDITIONS: Sarcopenia
Keywords: Neuromuscular electrical stimulation; Ageing; Protein ingestion
MeSH Terms: conditions — Sarcopenia | interventions — Dietary Proteins

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment during the day (Active Comparator): Neuromuscular electrical stimulation after a protein bolus, performed during the day
  Interventions: Procedure: Dietary protein plus NMES during the day
- Treatment prior to sleep (Active Comparator): Protein ingestion directly after one-legged NMES, directly prior to sleep
  Interventions: Procedure: Dietary protein plus NMES prior to sleep

INTERVENTIONS:
Procedure: Dietary protein plus NMES during the day — Neuromuscular electrical stimulation after a protein bolus, performed during the day
  Arms: Treatment during the day
Procedure: Dietary protein plus NMES prior to sleep — Neuromuscular electrical stimulation after a protein bolus, performed prior to sleep
  Arms: Treatment prior to sleep

SUMMARY:
In the present study, the effect of a bolus of intrinsically labeled milk directly after one-legged NMES (Neuromuscular Electrical Stimulation) will be studied under two conditions: during the day and prior to sleep

DETAILED DESCRIPTION:
In the present study, the effect of a bolus of intrinsically labeled milk directly after an hour of one-legged NMES (Neuromuscular Electrical Stimulation) will be studied under two conditions: during the day and immediately prior to sleep

ELIGIBILITY:
Inclusion Criteria:

* Age 65-85 years
* Male
* 18.5 ≤ BMI ≤ 30.0

Exclusion Criteria:

* Type II diabetes
* All co morbidities interacting with mobility and muscle metabolism of the lower limbs (e.g. arthrosis, arthritis, spasticity/rigidity, all neurological disorders, paralysis, hip/knee surgery).
* Use of anticoagulants, blood diseases, allergy for lidocaine
* Use of NSAIDs (non-steroidal anti-inflammatory drugs) and acetylsalicylic acid
* Patients suffering from PKU (Phenylketonuria)
* Presence of implantable cardioverter defibrillator and/or pacemaker
* Performed regular resistance type exercise in the past 6 months
* Use of any tools to assist during walking (cane/ crutches/ walker)
* (Partial) foot/ leg amputation

Ages: 65 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 16 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Incorporation of stable isotope amino acids into skeletal muscle tissue | 4-8 hours in the postprandial phase

SECONDARY OUTCOMES:
Plasma amino acid enrichment | 4-8 hours in the postprandial phase

CONTACTS AND LOCATIONS:
Overall Officials: Luc JC van Loon, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Centre +, Maastricht, Netherlands